CLINICAL TRIAL: NCT03777098
Title: Pilot Study of Strepic® Device for the Diagnosis of Group A Streptococcal Pharyngitis
Status: Completed | Type: Observational
Sponsor: David A. Talan (Other)
Collaborators: Light AI, Inc. (Unknown)
Responsible Party: Sponsor-Investigator, David A. Talan, Co-PI, Olive View-UCLA Education & Research Institute
Organization: Olive View-UCLA Education & Research Institute (Other)
Other Study IDs: 01-2018
Record Dates: First submitted 2018-12-11; First posted 2018-12-17 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Group A Streptococcal Infection
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Strepic® Device — The Strepic® device is a qualitative point-of-care diagnostic test for the detection of GAS pharyngitis. The test uses direct visualization of the pharynx with a light source of specified wavelengths, causing excitation of endogenous fluorophores that emit a characteristic colored light pattern. White light images may give additional diagnostic accuracy through use of an artificial intelligence analysis of a large set of images of GAS and non-GAS pharyngitis.

SUMMARY:
The objective of this pilot study is to acquire images using the Strepic® device, a clinical prototype that has been designed specifically as a viable, low-cost, commercially realizable autofluorescence-based diagnostic test, using (1) fluorescence and (2) white light image data, as well as other clinical data points. By acquiring and analyzing the images of pharyngeal bacterial fluorescence and white light patterns in patients with Group A Streptococcus (GAS)-associated pharyngitis and comparing them with those observed in non-GAS pharyngitis, it is believed an algorithm can be developed such that the device will improve the ability of clinicians to quickly and accurately identify GAS infections.

ELIGIBILITY:
Inclusion Criteria:

1. All patients aged 7-64 years of age with suspected GAS pharyngitis with modified Centor (McIsaac) score ≥2; and
2. Patient agrees to participate in study and patient or parent/guardian sign consent/assent form.

Exclusion Criteria:

1. Pharyngeal swab performed immediately prior to study team approach;
2. Prior enrollment in this study;
3. Pharyngeal symptoms >7 days;
4. Peritonsillar abscess;
5. Antibiotic use within one week of index visit;
6. Inability to open mouth to visualize the pharynx; and
7. Inability to understand English or Spanish, as study forms including consent and assent forms will be written in English and Spanish;
8. Woman who is pregnant (self-reported, pregnancy test will not be performed) or nursing;
9. Current prisoner (define as an individual involuntarily confined in a penal institution, including persons: (1) sentenced under a criminal or civil statue; (2) detained pending arraignment, trial, or sentencing; and (3) detained in other facilities (e.g., for drug detoxification or treatment of alcoholism) under statutes or commitment procedures providing such alternatives to criminal prosecution or incarceration in a penal institution).

Ages: 7 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients presenting to participating U.S. emergency departments or clinics with complaint of pharyngitis will be screened.
Sampling Method: Non-Probability Sample
Enrollment: 426 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Strepic Device Image | Day 1
  A picture of the participant's throat will be obtained at enrollment.
Throat culture or PCR result | Day 2
  The results of throat culture or PCR (depending on the site) will be recorded and compared to the Strepic Device image findings

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Moran, MD, Principal Investigator — Olive View-UCLA Education & Research Institute
Locations (1):
- Olive View-UCLA Medical Center, Sylmar, California, United States

IPD SHARING:
Plan to Share IPD: No